CLINICAL TRIAL: NCT00173498
Title: Common Allergens in Skin Tests for Adult Atopic Dermatitis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9461700672
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2005-09-15 (Estimated); Status verified 2005-07

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis, skin test
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
To analyze the common allergens revealed by skin tests in adult atopic dermatitis patients.

DETAILED DESCRIPTION:
The allergens involved in atopic patients are widely existed in our environment. Traditionally, we use serum specific IgE, skin prick test or intradermal test to verify the possible causative allergens in patients with atopic dermatitis. This study will evaluate the correlation between serum specific IgE, skin prick test, intradermal test, and patch test for common allergens in adult patients with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* patients with atopic dermatitis (according to Hanifin and Rajka criteria)
* age older than 16 years old

Exclusion Criteria:

* pregnancy

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60
Dates: Start 2005-07; Study Completion 2005-10

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Yu Chu, MD, Principal Investigator — Department of Dermatology, National Taiwan University Hospital
Locations (1):
- Department of Dermatology, National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Darsow U, Laifaoui J, Kerschenlohr K, Wollenberg A, Przybilla B, Wuthrich B, Borelli S Jr, Giusti F, Seidenari S, Drzimalla K, Simon D, Disch R, Borelli S, Devillers AC, Oranje AP, De Raeve L, Hachem JP, Dangoisse C, Blondeel A, Song M, Breuer K, Wulf A, Werfel T, Roul S, Taieb A, Bolhaar S, Bruijnzeel-Koomen C, Bronnimann M, Braathen LR, Didierlaurent A, Andre C, Ring J. The prevalence of positive reactions in the atopy patch test with aeroallergens and food allergens in subjects with atopic eczema: a European multicenter study. Allergy. 2004 Dec;59(12):1318-25. doi: 10.1111/j.1398-9995.2004.00556.x. PMID 15507101
- [Background] Ingordo V, Dalle Nogare R, Colecchia B, D'Andria C. Is the atopy patch test with house dust mites specific for atopic dermatitis? Dermatology. 2004;209(4):276-83. doi: 10.1159/000080848. PMID 15539888
- [Background] Weissenbacher S, Bacon T, Targett D, Behrendt H, Ring J, Darsow U. Atopy patch test--reproducibility and elicitation of itch in different application sites. Acta Derm Venereol. 2005;85(2):147-51. doi: 10.1080/00015550410024418. PMID 15823910